CLINICAL TRIAL: NCT07399717
Title: Assessing Role of Probiotics in Children Aged 6-36 Months Treated for Pneumonia at Phu Tho Provincial Obstetrics and Pediatrics Hospitals Within 2026-2027
Brief Title: Assessing Role of Probiotics in Children Aged 6-36 Months Treated for Pneumonia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anabio R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TNLS.2026.SNPT
Record Dates: First submitted 2026-01-16; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Pneumonia; Pneumonia in Children
Keywords: Acute respiratory infection; Adjunctive Treatment; Prevention; Nasal-oropharyngeal; Probiotic spray; Oral probiotic suspension; Bacillus spores; Children; Respiratory viruses; Bacterial co-infection
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Blinded, randomized, and controlled clinical trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: LiveSpo Navax and placebo 0.9% NaCl physiological saline are indistinguishable regarding taste and smell. The color and turbidity of LiveSpo Navax suspension are unrecognizable to investigators, trainers, child caregivers, children's parents, and children due to opaque plastic container. Similarly, LiveSpo Preg-Mom and oral reverse osmosis (RO) water were matched in sensory characteristics and packaging, thereby maintaining blinding of investigators, caregivers, parents, and participants.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): The placebo group receives 0.9% NaCl physiological saline. Caregivers will spray the children three times daily, administering 3 sprays in each nostril and 3 sprays in the throat each time (totally 6 sprays each time) for 8 weeks.
  The placebo group also receives oral Reverse Osmosis water twice daily, 5 mL per dose, for 8 weeks The Placebo group receives standard pneumonia treatment: oxygen (SpO2 < 92%) and antibiotics (ampicillin/sulbactam, with or without aminoglycosides/third-generation cephalosporins). Vancomycin/macrolides cover staphylococcal/atypical agents; levofloxacin is an alternate. Adjust per antibiogram. Supportive care: antipyretics, suctioning, fluids/electrolytes, nutrition, physiotherapy. Bronchodilators/corticosteroids are used for bronchospasm or severe pneumonia.
  Interventions: Other: Placebo
- Navax (Experimental): The Navax group receives LiveSpo® Navax product, which is NaCl 0.9% plus B. subtilis and B. clausii at 1 billion CFU/mL x 30 mL. Caregivers will spray the children three times daily, administering 3 sprays in each nostril and 3 in the throat, for 8 weeks.
  The Navax group also receives oral RO water twice daily, 5 mL per dose, for 8 weeks.
  The Navax group receives standard pneumonia treatment: oxygen (SpO2 < 92%) and antibiotics (ampicillin/sulbactam, with or without aminoglycosides/third-generation cephalosporins). Vancomycin/macrolides cover staphylococcal/atypical agents; levofloxacin is an alternate. Adjust per antibiogram. Supportive care: antipyretics, suctioning, fluids/electrolytes, nutrition, physiotherapy. Bronchodilators/corticosteroids are used for bronchospasm or severe pneumonia.
  Interventions: Combination Product: Navax
- Navax-PregMom (Experimental): The Navax-PregMom group receives LiveSpo® Navax product which is NaCl 0.9% plus B. subtilis and B. clausii at 1 billion CFU/mL x 30 mL. Caregivers will spray the children three times daily, administering 3 sprays in each nostril and 3 sprays in the throat each time for 8 weeks.
  The Navax-PregMom group is also given oral medication with LiveSpo® Preg-Mom which is RO water plus B. subtilis, B. clausii, and B. coagulans at 3 billion CFU/5mL. The children will receive the probiotic twice daily, with 1 vial per dosefor 8 weeks.
  The Navax-PregMom group receives standard pneumonia treatment: oxygen (SpO2 < 92%) and antibiotics (ampicillin/sulbactam, with or without aminoglycosides/third-generation cephalosporins). Vancomycin/macrolides cover staphylococcal/atypical agents; levofloxacin is an alternate. Adjust per antibiogram. Supportive care: antipyretics, suctioning, fluids/electrolytes, nutrition, physiotherapy. Bronchodilators/corticosteroids are used for bronchospasm or severe pneumonia.
  Interventions: Combination Product: Navax-PregMom

INTERVENTIONS:
Other: Placebo — 0.9% NaCl physiological saline is prepared by extracting 5 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B. Braun, Germany, product declaration No. Nasal-spraying 0.9% NaCl physiological saline is prepared by extracting 30 mL from 0.9% NaCl intravenous infusion 500 mL PP bottle (B.Braun, Germany, product declaration No. VD-32732-19), and then pouring it into the same opaque plastic spraying 20 mL-bottle that is used for nasal-oropharyngeal probiotic spray.
  Reverse Osmosis water (Aquafina, PepsiCo) is produced under ISO 9001:2015 and ISO 22000:2018 standards. The RO water ampoules are produced using a similar process as the LIVESPO PREG-MOM but contain 5 mL of high-quality RO water from Aquafina.
  Arms: Placebo
Combination Product: Navax — In Vietnam, LiveSpo Navax is manufactured as a Class-A medical device (Product declaration: No. 210001337/PCBA-HN) in accordance with manufacturing standards approved by the Hanoi Health Department, Ministry of Health, Vietnam (Certificate No. YT117-19), and ISO 13485:2016. LiveSpo Navax product is prepared in the form of NaCl 0.9% plus B. subtilis and B. clausii at 1 billion CFU/mL x 20 mL.
  RO water (Aquafina, PepsiCo) produced under ISO 9001:2015 and ISO 22000:2018 standards. The RO water ampoules are produced using a similar process as the LIVESPO PREG-MOM but contain 5 mL of high-quality RO water from Aquafina.
  Arms: Navax
Combination Product: Navax-PregMom — In Vietnam, LiveSpo Navax is manufactured as a Class-A medical device (Product declaration: No. 210001337/PCBA-HN) in accordance with manufacturing standards approved by the Hanoi Health Department, Ministry of Health, Vietnam (Certificate No. YT117-19), and ISO 13485:2016. LiveSpo Navax product is prepared in the form of NaCl 0.9% plus B. subtilis and B. clausii at 1 billion CFU/mL x 30 mL.
  LiveSpo PREG-MOM has a registration number 7695/2020/ĐKSP issued by the Food Safety Department of the Ministry of Health in Vietnam.
  Arms: Navax-PregMom

SUMMARY:
The main questions this study aims to answer are:

* Does using probiotic nasal spray (LiveSpo Navax containing Bacillus subtilis and Bacillus clausii, 1x10^9 CFU/mL), with or without oral probiotics (LiveSpo Pregmom containing Bacillus subtilis, Bacillus clausii, and Bacillus coagulans, 3x10^9 CFU/5 mL), help children recover better from pneumonia when added to standard medical treatment?
* Does using these adjunctive probiotics support reduce the recurrence of respiratory and gastrointestinal symptoms after hospital discharge? Researchers will compare three groups of children to see whether probiotic nasal spray alone or probiotic nasal spray combined with oral probiotics works better than placebo.

All participants will receive standard medical treatment for pneumonia. In addition, they will be randomly assigned to one of three study groups to receive adjunctive probiotic support in 2 months:

* Control group: receives a saline nasal-throat spray (0.9% NaCl) and oral placebo liquid (RO water).
* Nasal probiotic group: receives a probiotic LiveSpo® Navax nasal-throat spray and oral placebo liquid (RO water).
* Nasal plus oral probiotic group: receives a probiotic LiveSpo® Navax nasal-throat spray plus LiveSpo® Preg-Mom oral probiotic suspension.

Participants will:

* Use a nasal-throat spray three times a day.
* Take an oral liquid twice daily.
* Start using the study products during their hospital stay and continue for 8 weeks (2 months) from admission.
* Be followed by the study team during hospitalization and at Day 30 and Day 60 after admission. The probiotic and placebo products look, smell, and taste the same so that neither the parents nor the study staff know which product each child receives.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled clinical trial conducted at Phu Tho Provincial Obstetrics and Pediatrics Hospital to evaluate Bacillus spore probiotics delivered by nasal-oropharyngeal spray (LiveSpo® Navax) with or without an oral probiotic suspension (LiveSpo® Preg-Mom) as an adjunct to standard medical treatment in children aged 6-36 months hospitalized with pneumonia.

A total of 330 eligible children will be randomly assigned in a 1:1:1 ratio into three groups (n = 110 per group):

the Control group receiving 0.9% sodium chloride nasal-oropharyngeal spray and oral RO water, the Navax group receiving Bacillus spore probiotic nasal-oropharyngeal spray and oral RO water, and the Navax-PregMom group receiving Bacillus spore probiotics both as nasal spray and oral suspension. All participants receive standard-of-care treatment according to hospital guidelines, with differences between groups limited to the assigned study interventions.

The nasal-oropharyngeal spray is administered as three sprays per nostril and throat per dose, three times daily, and the oral intervention is administered at a daily dose of 5 mL, twice daily. Interventions are initiated during hospitalization and continued for up to two months from admission.

Rationale and need: Pediatric pneumonia often proceeds upper-airway infection and is characterized by pathogen colonization of-and inflammation within the naso-/oropharyngeal mucosa. Accordingly, a nasal-throat Bacillus spore spray could serve as a local adjunct to maintain airway hygiene and mucosal restitution while potentially mitigating the load of respiratory viruses and bacterial co-pathogens at the site of infection. Concomitant interventions for hospitalized children with pneumonia, including supportive care and administration of medications (such as antibiotics), could perturb the gut microbiota and lead to gastrointestinal symptoms before or after treatment. An oral Bacillus spore suspension is expected to complement the local intervention by acting through the gut-immune interface, thereby supporting systemic immune modulation and recovery beyond the upper airway.

Crucially, most of the available clinical trials examine probiotics as monotherapy (e.g., oral or nasal alone), and did not sufficiently address outcomes related to combining both routes in the same treatment. The purpose of this trial is to directly examine the hypothesis that there will be an additive effect of providing concurrent Bacillus nasally (B. subtilis ANA4 + B. clausii ANA39) and orally (B. subtilis ANA46 + B. clausii ANA39 + B. coagulans ANA40) administered probiotics in hospitalized children with pneumonia. The expected mechanism is that the combined regimen may better support treatment and prevention of recurrence by reducing viral load, bacterial co-infection, and pro-inflammatory cytokines, while improving nasal and gut microbiota profiles.

After written informed consent is obtained, baseline demographic and clinical data are collected using standardized questionnaires and medical records.

During inpatient treatment, physicians and nurses monitor and record daily clinical symptoms, including fever, cough, tachypnea, chest indrawing, wheezing, crackles, and gastrointestinal manifestations, as well as length of hospital stay and use of medications such as antibiotics, antiviral agents, and supportive therapies. Nasopharyngeal, blood and stool samples are collected at predefined time points according to the protocol (mandatory at day 0 and day 3, and optional at day 30 and day 60). All of these samples are processed to quantify inflammatory cytokines (IL-6, IL-8, IL-10, IL-17, IL-23, TNF-α) and IgA using ELISA, and to detect respiratory viruses, bacterial co-pathogens, and B. subtilis, B. clausii, and B. coagulans by real-time PCR. Stratified subsamples of stool and nasopharyngeal samples (n = 15-20 per group x 2 time points) undergo 16S rRNA gene sequencing to assess changes in respiratory (at day 30 vs. day 0) and gut microbiota (at day 30 vs. day 0) diversity and taxonomic composition. After discharge, children are followed up at day 30 and/or day 60 through outpatient visits or structured interviews with parents or caregivers to document recurrence of respiratory or gastrointestinal symptoms, rehospitalization, and post-discharge medication use. Parents or caregivers are instructed not to administer other probiotic products (except yoghurt) or Bacillus spore nasal preparations during the study period.

All medical records are collected, scanned, and stored in electronic format. Patient data are systematically organized into databases for analysis. Reduction in pathogen load is assessed by comparing real-time PCR cycle threshold (Ct) values at discharge or follow-up with baseline using the 2^-ΔCt method. Changes in cytokine and IgA concentrations are evaluated by comparing median values before and after intervention. The presence of B. subtilis, B. clausii, and B. coagulans in samples is expressed using Ct values from TaqMan probe assays. Statistical analyses and graphical presentations are performed using GraphPad Prism (version 10.2.3), IBM SPSS Statistics (version 27), and R software (version 4.4.2), with a two-sided significance level set at p < 0.05. Randomization and double blinding are applied to minimize random and systematic bias, and treatment allocation codes remain concealed until completion of data analysis, except in cases of serious adverse events requiring emergency unblinding.

ELIGIBILITY:
Inclusion Criteria:

* Children (male/female) aged 6-36 months diagnosed and hospitalized for treatment for pneumonia.
* Parents or guradians of the children agree to participate in the study, explain, and sign the research consent form.

Exclusion Criteria:

* Children who need ventilator support.
* Children who have had rhinoplasty surgery, nasal ulcers, nasal polyps or any nasal deformity that affects the use of the study product.
* Children who get transferred or leave the treatment unit (not for professional reasons).
* Children who have experienced congenital immunodeficiency or infectious disease (eg, HIV).
* Children who are concurrently participating in another clinical trial or participated in a clinical trial within 30 days before selection.
* Children who are under long-term medication (more than 7 consecutive days) within 30 days before selection.
* Children with allergy or hypersensitivity to any ingredient of the study product.

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Estimated)
Dates: Start 2026-01-26 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Number of days with typical clinical symptoms of pneumonia | Daily assessments will be conducted during hospitalization, from admission (Day 0) through discharge. The duration of hospitalization is variable, averaging 10 days.
  Symptoms to be assessed include fever, cough, tachypnea, chest retraction, wheezing, crackles, moist rales, diarrhea, etc.
Number of days of inpatient treatment | Daily assessments will be conducted during hospitalization, from admission (Day 0) through discharge. The duration of hospitalization is variable, averaging 10 days.
  The total number of days a participant stays in the hospital for treatment during the study period.

SECONDARY OUTCOMES:
Use of medications and supportive treatments during hospitalization | Daily assessments will be conducted during hospitalization, from admission (Day 0) through discharge. The duration of hospitalization is variable, averaging 10 days.
  Percentage of children using various medications (antiviral, antibiotics, and other symptomatic treatments such as antipyretics, anti-inflammatory drugs, anti-allergics, etc.) and supportive treatments (oxygen therapy, nebulization, etc.) throughout the inpatient treatment period, including the starting date of use, type of medication, and total number of days used.
Inflammatory cytokine and IgA levels in clinical samples | Days 0 and 3 (mandatory), and on discharge days 30 and 60 (optional)
  Cytokine concentrations, including IL-6 (pg/mL), IL-8 (pg/mL), TNF-α (pg/mL), Immunoglobulin A (IgA) (µg/mL) in nasopharyngeal swabs, IL-10 (pg/mL), IL-17 (pg/mL), IL-23 (pg/mL) in blood, will be measured using ELISA.
Presence of probiotic bacterial spores | Days 0 and 3 (mandatory), and on discharge days 30 and 60 (optional)
  Presence of beneficial bacterial spores B. subtilis, B. clausii, and B. coagulans in nasopharyngeal swabs and samples measured using Real-time PCR
Semi-quantitative changes in respiratory viral and bacterial pathogen loads | Days 0 and 3 (mandatory), and on discharge days 30 and 60 (optional)
  Semi-quantitative changes in loads of several common respiratory pathogens, including at least 3 of 6 common viruses (1) RSV, (2) influenza A-B, (3) rhinovirus, (4) adenovirus, (5) parainfluenza virus, (6) Covid-19, and 3 common bacterial co-infections (1) S. pneumoniae, (2) H. influenzae, and (3) Moraxella cattaralis
Proportion of children with diarrheal symptoms during hospitalization | Daily assessments will occur during hospitalization, from admission (Day 0) until discharge. The duration of hospitalization is variable, averaging 10 days.
  The proportion of children with diarrheal symptoms during hospital stay: having more than three bowel movements per day, with loose or watery stools, corresponding to Bristol Stool Form Scale (BSFS) types 5-7, with or without visible mucus in the stool
Recurrence of acute respiratory and gastrointestinal symptoms | Day 30 and/or day 60 of the study
  The recurrence rate of acute respiratory and gastrointestinal symptoms recorded through follow-up visits or interviews with parents/guardians
Hospital readmission due to respiratory and gastrointestinal illnesses | Day 30 and/or day 60 of the study
  The rate of readmission due to respiratory and gastrointestinal illnesses at the follow-up time points recorded through follow-up visits or interviews with parents/guardians
Use of Medications During Follow-up | Day 30 and/or day 60 of the study
  The rate of children using antiviral drugs, antibiotics, and other symptomatic treatments such as antipyretics, anti-inflammatory drugs, anti-allergics, etc. recorded through follow-up visits or interviews with parents/guardians
IgA levels in stool samples | Time Frame: Days 0 and 3 (mandatory), and on discharge days 30 and 60 (optional)
  Immunoglobulin A (IgA) (µg/g) in stool will be measured using ELISA.

OTHER OUTCOMES:
Changes in nasal microbiota composition and diversity | Day 0 and one of follow-up time points Day 3, 30, or 60
  Changes in nasal microbiota, analysis of alpha, beta, phylum, family, genus, and species diversity changes using 16S rRNA NGS technique (V3-V4 region), in nasopharyngeal swab samples
Changes in gut microbiota composition and diversity | Day 0 and one of follow-up time points Day 3, 30, or 60
  Changes in gut microbiota, analysis of alpha, beta, phylum, family, genus, and species diversity changes using 16S rRNA NGS technique (V3-V4 region), in stool samples

CONTACTS AND LOCATIONS:
Overall Officials: Loc V Nguyen, MD., Principal Investigator — Phu Tho Provincial Obstetrics and Pediatrics Hospitals; Anh TV Nguyen, Assoc. Prof, Study Chair — Spobio Research Center, Anabio R&D
Locations (1):
- Phu Tho Provincial Obstetrics and Pediatrics Hospitals, Phú Thọ, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Data or samples share that will be coded, with no PHI include. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research and will be provided following review and approval of a study protocol, informed consent form (ICF), and clinical study reports (CSR). For more information or to submit a request, please contact anabio.rd2021@gmail.com

REFERENCES:
- [Background] Dao BN, Le HDT, Ta TB, et al. Relationship between serum TNF-α, IL-6, and IL-10 levels and disease severity, and changes in the cytokines after treatment in patients with bacterial community-acquired pneumonia. Pneumon. 2023; doi.org/10.18332/pne/170181
- [Background] Zhang Z, Dou H, Tu P, Shi D, Wei R, Wan R, Jia C, Ning L, Wang D, Li J, Dong Y, Xin D, Xu B. Serum cytokine profiling reveals different immune response patterns during general and severe Mycoplasma pneumoniae pneumonia. Front Immunol. 2022 Dec 22;13:1088725. doi: 10.3389/fimmu.2022.1088725. PMID: 36618370; PMCID: PMC9813340.
- [Background] Ness-Cochinwala M, Totapally BR. A Comprehensive Review of Pediatric Necrotizing Pneumonia. Children. 2025; 12(9):1248. doi.org/10.3390/children12091248
- [Background] Roh EJ, Shim JY, Chung EH. Epidemiology and surveillance implications of community-acquired pneumonia in children. Clin Exp Pediatr. 2022 Dec;65(12):563-573. doi: 10.3345/cep.2022.00374. Epub 2022 Oct 17. PMID: 36265520; PMCID: PMC9742763.
- [Background] Turalde-Mapili MWR, Mapili JAL, Turalde CWR, Pagcatipunan MR. The efficacy and safety of nirsevimab for the prevention of RSV infection among infants: A systematic review and meta-analysis. Front Pediatr. 2023 Apr 4;11:1132740. doi: 10.3389/fped.2023.1132740. PMID: 37082704; PMCID: PMC10110918.
- [Background] Han JS, Jang SH, Jeon JS, Lee KB, Kim JK. Epidemiological Shifts in Respiratory Virus Infections Among Older Adults (≥65 Years) Before and After the COVID-19 Pandemic: An 18-Year Retrospective Study in the Republic of Korea. Microorganisms. 2025 Oct 3;13(10):2301. doi: 10.3390/microorganisms13102301. PMID: 41156761; PMCID: PMC12566155.
- [Background] Khieu, T.H., Le, D.P., Nguyen, B.T. et al. Alleviating symptoms of paediatric acute rhinosinusitis and acute otitis media with otorrhea using nasal-spraying Bacillus probiotics: a randomized controlled trial. Sci Rep 15, 3410 (2025). https://doi.org/10.1038/s41598-025-87372-2
- [Background] Zou, Y., Huang, F., Sun, J. et al. The role of IFN-γ/CXCL10 axis in Mycoplasma pneumonia infection. Sci Rep 15, 2671 (2025). https://doi.org/10.1038/s41598-024-84969-x
- [Background] Chen Z, Liu Y, Huang W. Alveolar macrophage modulation via the gut-lung axis in lung diseases. Front Immunol. 2023 Nov 21;14:1279677. doi: 10.3389/fimmu.2023.1279677. PMID: 38077401; PMCID: PMC10702770.
- [Background] Thi Le, H., Thi Bich Phung, T., Thi Bui, H. et al. Nasal-spraying Bacillus spore probiotics for pneumonia in children with respiratory syncytial virus and bacterial co-infections: a randomized clinical trial. Commun Med 5, 336 (2025). https://doi.org/10.1038/s43856-025-01029-9
- [Background] Tran, X.D., Hoang, VT., Goumballa, N. et al. Viral and bacterial microorganisms in Vietnamese children with severe and non-severe pneumonia. Sci Rep 14, 120 (2024). https://doi.org/10.1038/s41598-023-50657-5
- [Background] Tran, D.M., Tran, T.T., Phung, T.T.B. et al. Nasal-spraying Bacillus spores as an effective symptomatic treatment for children with acute respiratory syncytial virus infection. Sci Rep 12, 12402 (2022). https://doi.org/10.1038/s41598-022-16136-z